CLINICAL TRIAL: NCT01936324
Title: A Study of the Safety, Tolerability and Preliminary Efficacy of DRM01B Topical Gel in Healthy Volunteers and Subjects With Acne Vulgaris
Brief Title: A Safety, Tolerability and Preliminary Efficacy Study of DRM01B Topical Gel
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dermira, Inc. (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRM01B-ACN01
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 1 (Experimental): Olumacostat Glasaretil Gel, 7.5%, applied twice daily to the face for 7 days in healthy volunteers
  Interventions: Drug: Olumacostat Glasaretil Gel, 7.5%
- Phase 2a (Experimental): Olumacostat Glasaretil Gel, 7.5%, or Olumacostat Glasaretil Gel, Vehicle, applied twice daily to the face for 12 weeks
  Interventions: Drug: Olumacostat Glasaretil Gel, 7.5%; Other: Olumacostat Glasaretil Gel, Vehicle

INTERVENTIONS:
Drug: Olumacostat Glasaretil Gel, 7.5% — Gel containing Olumacostat Glasaretil
  Other Names: DRM01
Other: Olumacostat Glasaretil Gel, Vehicle — Vehicle (placebo) gel
  Arms: Phase 2a

SUMMARY:
This is a Phase 1/2a study.

The purpose of Phase 1 was to evaluate the safety and tolerability of DRM01B Topical Gel in 6 healthy volunteers.

The purpose of Phase 2a was to assess the safety, tolerability and preliminary efficacy of DRM01B Topical Gel compared to vehicle in subjects with acne vulgaris on the face.

ELIGIBILITY:
Phase 1 Inclusion Criteria

1. Signed informed consent
2. Willing to comply with the requirements of the protocol
3. Males or non-pregnant, non-lactating females
4. Age ≥ 18 years
5. Was in good health and free from any clinically significant disease, as determined by the investigator
6. If female and of childbearing potential, was willing to use an accepted method of birth control during study participation and for 30 days after the last application of study drug. Females were considered to be of childbearing potential unless they had been surgically sterilized (hysterectomy, bilateral oophorectomy, tubal ligation), had been diagnosed as infertile, had a same-sex partner or vasectomized male partner, were postmenopausal for at least 1 year, or were abstinent. Acceptable methods of birth control were defined as: abstinence, oral contraceptives, contraceptive patches/implants; Depo-Provera®, double barrier methods (e.g., condom and spermicide) or an intrauterine device (IUD). The birth control method must have been stable/unchanged for 30 days prior to baseline.
7. If male, was vasectomized or agreed to use an accepted method of birth control with female partner during study participation and for 30 days after the last application of study drug.

Phase 1 Exclusion Criteria

1. Females who were pregnant, planning to become pregnant during the course of the study, or were breast-feeding
2. Had a known hypersensitivity to DRM01B or its excipients
3. Had any skin condition that may have interfered with the safety evaluations during the study
4. Had a clinical chemistry or hematology laboratory value at screening that was considered clinically significant, in the opinion of the investigator
5. Participated in an investigational drug study within 30 days prior to screening
6. Were considered a poor medical risk because of other systemic diseases or active uncontrolled infections, in the opinion of the investigator. Any other condition which, in the judgment of the investigator, would put the subject at unacceptable risk for participation in the study.

Phase 2a Inclusion Criteria

1. Signed informed consent
2. Willing to comply with the requirements of the protocol
3. Male or non-pregnant, non-lactating females
4. Age ≥ 18 years
5. If female and of childbearing potential, was willing to use an accepted method of birth control during study participation and for 30 days after the last study drug application. Females were considered to be of childbearing potential unless surgically sterilized (hysterectomy, bilateral oophorectomy, tubal ligation), had been diagnosed as infertile, had same sex partner or vasectomized male partner, or were postmenopausal for at least 1 year. Acceptable methods of birth control were defined as: abstinence, oral contraceptives, contraceptive patches/implants; Depo-Provera®, double barrier methods (e.g., condom and spermicide) or an IUD. The birth control method must have been stable/unchanged for 12 weeks prior to baseline and must have remained unchanged during study participation.
6. If male, was vasectomized or agreed to use an accepted method of birth control with female partner during study participation and for 30 days after the last study drug application.
7. Subjects were in good health and free from any disease that, in the opinion of the investigator, would have put the subject at risk during participation in the study.
8. Clinical diagnosis of facial acne vulgaris defined as:

   * At least 20 inflammatory lesions
   * At least 20 noninflammatory lesions
   * IGA of 3 or greater
9. Willing to refrain from using any treatments, other than the investigational product, including antibiotics, for acne present on the face. Topical acne treatments that did not have significant or measurable systemic absorption (e.g., benzoyl peroxide, salicylic acid) were allowed for treatment of acne of the back, shoulders, and chest only.

Phase 2a Exclusion Criteria

1. Females who were pregnant, planning to become pregnant during the course of the study, or breast-feeding
2. Had a known hypersensitivity to DRM01B or its excipients
3. Had any skin condition that may have interfered with evaluation of safety or acne vulgaris (e.g., rosacea; seborrheic dermatitis; perioral dermatitis; corticosteroid-induced acne or folliculitis)
4. Had excessive facial hair that would have interfered with diagnosis or assessment of acne vulgaris
5. Had excessive sun exposure, in the opinion of the investigator, or use of tanning booths
6. Had active cystic acne or acne conglobata, acne fulminans, and secondary acne
7. Had 2 or more active nodular lesions
8. Had a clinical chemistry or hematology laboratory value at screening that was considered clinically significant, in the opinion of the investigator
9. Participated in an investigational drug study within 30 days prior to screening
10. Subjects who were a poor medical risk because of other systemic diseases or active uncontrolled infections, in the opinion of the investigator
11. Any other condition that, in the judgment of the investigator, would have put the subject at unacceptable risk during participation in the study
12. Treatment with over-the-counter (OTC) topical medications for the treatment of acne vulgaris including benzoyl peroxide, topical anti-inflammatory medications, corticosteroids, α-hydroxy/glycolic acid on the face within 2 weeks prior to baseline
13. Treatment with systemic corticosteroids within 4 weeks prior to baseline (Note: use of intranasal and inhaled corticosteroids was allowed for seasonal allergies and asthma)
14. Treatment with systemic antibiotics, systemic anti-acne drugs, or systemic anti-inflammatory drugs within 4 weeks prior to baseline
15. Prescription topical retinoid use on the face within 4 weeks of baseline (e.g., tretinoin, tazarotene, adapalene).
16. Treatment with a new hormonal therapy or dose change to an existing hormonal therapy within 12 weeks prior to baseline. The dose and frequency of use of any hormonal therapy started more than 12 weeks prior to baseline must have remained unchanged throughout the study. Hormonal therapies included, but were not limited to, estrogenic and progestational agents, such as birth control pills.
17. Prior use of androgen receptor blockers (such as spironolactone or flutamide)
18. Oral retinoid use (e.g., isotretinoin) within 12 months prior to baseline or vitamin A supplements greater than 10,000 units/day within 6 months of baseline
19. Facial procedures (chemical or laser peel, microdermabrasion, etc.) within the past 8 weeks or during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice Drew, Study Director — Dermira, Inc.
Locations (12):
- Canada (12):
  - Guildford Dermatology Specialist Inc, Surrey, British Columbia
  - Ultranova Skincare, Barrie, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - Institute of Cosmetic & Laser Surgery, Oakville, Ontario
  - Skin Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - Research Toronto, Toronto, Ontario
  - K. Papp Clinical Research Inc., Waterloo, Ontario
  - Windsor Clinical Research, Inc., Windsor, Ontario
  - Innovaderm Research, Inc, Montreal, Quebec
  - Siena Medical Research, Montreal, Quebec
  - Centre de Recherche Dermetologique du Quebec Metropolitain (CRDQ), Québec

RESULTS

PARTICIPANT FLOW:
Groups:
- Olumacostat Glasaretil Gel, 7.5%, Phase 1: Olumacostat Glasaretil Gel, 7.5%, applied twice daily to the face for 7 days in healthy volunteers
- Olumacostat Glasaretil Gel, 7.5%, Phase 2a: Olumacostat Glasaretil Gel, 7.5%, applied twice daily to the face for 12 weeks
- Olumacostat Glasaretil Gel, Vehicle, Phase 2a: Olumacostat Glasaretil Gel, Vehicle, applied twice daily to the face for 12 weeks
Period: Overall Study
Arm/Group | Olumacostat Glasaretil Gel, 7.5%, Phase 1 | Olumacostat Glasaretil Gel, 7.5%, Phase 2a | Olumacostat Glasaretil Gel, Vehicle, Phase 2a
Started | 6 | 53 | 55
Completed | 6 | 47 | 50
Not Completed | 0 | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olumacostat Glasaretil Gel, 7.5%, Phase 1 | Olumacostat Glasaretil Gel, 7.5%, Phase 2a | Olumacostat Glasaretil Gel, Vehicle, Phase 2a | Total
Number analyzed (Participants) | 6 | 53 | 55 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 12 | 12 | 24
  Between 18 and 65 years | 6 | 41 | 43 | 90
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (11.3) | 23.9 (6.1) | 26.5 (9.0) | 26.0 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 33 | 38 | 73
  Male | 4 | 20 | 17 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 3 | 8
  Not Hispanic or Latino | 6 | 48 | 52 | 106
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 1 | 4
  Asian | 0 | 9 | 10 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 6 | 5 | 11
  White | 5 | 33 | 38 | 76
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 6 | 53 | 55 | 114
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick Skin Type is a scale to numerically classify skin color, defined by the response to ultraviolet (UV) light with the following categories:
  Type I Burns easily, rarely tans Type II Burns easily, tans minimally Type III Burns moderately, tans gradually Type IV Burns minimally, tans well Type V Rarely burns, tans profusely Type VI Never burns, deeply pigmented
  Participants
    Type I | 0 | 3 | 3 | 6
    Type II | 2 | 8 | 14 | 24
    Type III | 3 | 18 | 18 | 39
    Type IV | 1 | 16 | 13 | 30
    Type V | 0 | 3 | 2 | 5
    Type VI | 0 | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean Absolute Change in Acne Lesion Counts (Inflammatory) From Baseline to Week 12 in Phase 2a
Description: Mean absolute change in acne lesion counts (inflammatory) from baseline to Week 12 in Phase 2a
Time Frame: Baseline and Week 12
Population: Intent-to-Treat
Measure: Least Squares Mean (Standard Error); unit: Lesions
Arm/Group | Olumacostat Glasaretil Gel, 7.5%, Phase 2a | Olumacostat Glasaretil Gel, Vehicle, Phase 2a
Number analyzed (Participants) | 53 | 55
Lesions | -19.865 (1.107) | -14.296 (1.079)
Statistical Analysis 1: Comparison: Olumacostat Glasaretil Gel, 7.5%, Phase 2a vs Olumacostat Glasaretil Gel, Vehicle, Phase 2a; Test type: Other; p = 0.0003, ANCOVA; ANCOVA model with terms of treatment, baseline lesion count, and center

2. Primary Outcome: Mean Absolute Change in Acne Lesion Counts (Non-inflammatory) From Baseline to Week 12 in Phase 2a
Description: Mean absolute change in acne lesion counts (non-inflammatory) from baseline to Week 12 in Phase 2a
Time Frame: Baseline and Week 12
Population: Intent-to-Treat
Measure: Least Squares Mean (Standard Error); unit: Lesions
Arm/Group | Olumacostat Glasaretil Gel, 7.5%, Phase 2a | Olumacostat Glasaretil Gel, Vehicle, Phase 2a
Number analyzed (Participants) | 53 | 55
Lesions | -20.131 (1.902) | -12.357 (1.856)
Statistical Analysis 1: Comparison: Olumacostat Glasaretil Gel, 7.5%, Phase 2a vs Olumacostat Glasaretil Gel, Vehicle, Phase 2a; Test type: Other; p = 0.0032, ANCOVA; ANCOVA model with terms of treatment, baseline lesion count, and center

3. Primary Outcome: Percentage of Subjects Who Achieved ≥ 2-grade Improvement in the Investigator Global Assessment of Acne (IGA) From Baseline to Week 12 in Phase 2a
Description: Percentage of subjects who achieved ≥ 2-grade improvement in the investigator global assessment of acne (IGA) from baseline to Week 12 in Phase 2a
  Scoring Criteria for Investigator Global Assessment 0 - Clear skin with no inflammatory or noninflammatory lesions
  1. - Almost clear; rare noninflammatory lesions with no more than one small inflammatory lesion
  2. - Mild severity; greater than Grade 1; some noninflammatory lesions with no more than a few inflammatory lesions (papules/pustules only, no nodular lesions)
  3. - Moderate severity; greater than Grade 2; up to many noninflammatory lesions and may have some inflammatory lesions, but no more than one small nodular lesion
  4. - Severe; greater than Grade 3; up to many noninflammatory and inflammatory lesions, but no more than a few nodular lesions
Time Frame: Baseline and Week 12
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Olumacostat Glasaretil Gel, 7.5%, Phase 2a | Olumacostat Glasaretil Gel, Vehicle, Phase 2a
Number analyzed (Participants) | 53 | 55
Participants
  Success | 13 | 4
  Failure | 40 | 51
Statistical Analysis 1: Comparison: Olumacostat Glasaretil Gel, 7.5%, Phase 2a vs Olumacostat Glasaretil Gel, Vehicle, Phase 2a; Test type: Other; p = 0.0070, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by study center

ADVERSE EVENTS:
Time Frame: Baseline to Week 12
Description: The Total Participants at risk are based on the Safety Population defined as Participants who were randomized and received at least one confirmed dose of study drug.
Arm/Group | Olumacostat Glasaretil Gel, 7.5%, Phase 1 | Olumacostat Glasaretil Gel, 7.5%, Phase 2a | Olumacostat Glasaretil Gel, Vehicle, Phase 2a
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/53 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/53 | 1/55
Other Adverse Events (participants affected / at risk) | 0/6 | 29/53 | 17/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olumacostat Glasaretil Gel, 7.5%, Phase 1 (N=6) | Olumacostat Glasaretil Gel, 7.5%, Phase 2a (N=53) | Olumacostat Glasaretil Gel, Vehicle, Phase 2a (N=55)
Ankle Fracture Right (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olumacostat Glasaretil Gel, 7.5%, Phase 1 (N=6) | Olumacostat Glasaretil Gel, 7.5%, Phase 2a (N=53) | Olumacostat Glasaretil Gel, Vehicle, Phase 2a (N=55)
Application site dryness (General disorders) | 0 | 4 | 3
Application site erythema (General disorders) | 0 | 4 | 0
Application site pain (General disorders) | 0 | 4 | 3
Gastroenteritis (Infections and infestations) | 0 | 3 | 1
Nasopharyngitis (Infections and infestations) | 0 | 13 | 7
Headache (Nervous system disorders) | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes